CLINICAL TRIAL: NCT00931216
Title: Integration of HIV Care and Treatment Into Antenatal Care in Migori District, Kenya
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); Kenya Medical Research Institute (Other)
Responsible Party: Principal Investigator, Craig Cohen, Professor, University of California, San Francisco
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: KE.07.0055
Record Dates: First submitted 2009-06-30; First posted 2009-07-02 (Estimated); Last update posted 2012-04-10 (Estimated); Status verified 2012-04

CONDITIONS: HIV Infections
Keywords: PMTCT; Vertical transmission of HIV; Pregnant women; Infant HIV testing; Kenya; AIDS
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Integrated ANC, PMTCT and HIV Services (Experimental): HIV care and treatment services are integrated into antenatal care (ANC) services for women testing positive within the ANC at this facility.
  Interventions: Procedure: Integrated ANC, PMTCT, HIV services
- Non-Integrated Services (No Intervention): Women testing positive in the ANC department are referred for care at the HIV clinic. HIV care and treatment services are not provided within the ANC at facilities randomized to this arm.

INTERVENTIONS:
Procedure: Integrated ANC, PMTCT, HIV services — Of the 12 study clinics, 6 will be randomized to receive the intervention. At these 6 facilities, health care providers within the ANC department will be trained to also provide HIV/PMTCT care. Women testing positive within ANC clinics at integrated facilities will receive ANC, PMTCT and HIV services within the same visit/same service provider rather than being referred for HIV care and treatment.
  Arms: Integrated ANC, PMTCT and HIV Services

SUMMARY:
This study seeks to determine the most effective way to reach and provide pregnant women with accessible, comprehensive, and high quality HIV care and treatment.

DETAILED DESCRIPTION:
This study uses a prospective cluster randomized design. Twelve clinics similar in size, population, and services in Migori district, Kenya that provide ANC have been randomly assigned to receive "integrated ANC, PMTCT & HIV services" (intervention arm) or "non-integrated services" (control arm). At the intervention clinics, pregnant women will receive ANC, PMTCT and HIV care and treatment (including HAART if required) at the same clinic visit from the ANC provider. At the control clinics, women will receive antenatal care and PMTCT services with referral to the HIV care and treatment department located in the same facility. The control sites more closely resemble the current approach followed for care and treatment of HIV-infected pregnant women in Kenya. The content of ANC, PMTCT, and HIV care will be the same in the two study arms and will follow current Kenyan national guidelines. The only difference between the two arms will be the provider/location of HIV care and treatment.

Outcomes will be compared for HIV-positive pregnant women who attend intervention versus control facilities. In addition we will conduct qualitative research with health care providers at the study health facilities in order to learn provider perspectives on the two service models and to explore the effects of integration on provider job satisfaction (including work load).

ELIGIBILITY:
Inclusion Criteria:

* FOR SITE INCLUSION:

  * Each site must provide ANC services
  * Each site must provide HIV testing services for pregnant women
  * Each site must have an average of at least 20 new ANC clients per month
* FOR ENROLLMENT OF HIV-POSITIVE WOMEN:

  * All women testing HIV-positive at one of the 12 ANC clinics included in the study will be asked to participate in the study
* FOR HEALTH PROVIDER INCLUSION IN INTERVIEWS:

  * Health care staff must work within the ANC clinic at selected facilities
  * Staff must be able to read and speak English well enough to complete the informed consent process, participate in a one-on-one in-depth interview in English and complete a brief self-administered questionnaire

Exclusion Criteria:

* FOR SITE EXCLUSION:

  * If all of inclusion criteria are not met the site will be excluded
  * If site is already providing integrated ANC/HIV care services
* FOR HEALTH PROVIDER INCLUSION IN INTERVIEWS:

  * If all of inclusion criteria are not met the site will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1172 (Actual)
Dates: Start 2009-06; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Vertical transmission of HIV | 3 months postpartum

SECONDARY OUTCOMES:
Maternal HIV treatment outcomes | 6 months, 1 year
Provider job satisfaction | 1 year
Infant HIV testing uptake | 3 months postpartum
Patient enrollment, retention and adherence in HIV care and treatment | 6 months, 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Craig R Cohen, MD, MPH, Principal Investigator — University of California, San Francisco; Janet M Turan, PhD, MPH, Study Director — University of California, San Francisco; Elizabeth A Bukusi, MBChB, PhD, Principal Investigator — Kenya Medical Research Institute
Locations (1):
- Migori District Hospital, Migori, Kenya

REFERENCES:
- [Derived] Turan JM, Steinfeld RL, Onono M, Bukusi EA, Woods M, Shade SB, Washington S, Marima R, Penner J, Ackers ML, Mbori-Ngacha D, Cohen CR. The study of HIV and antenatal care integration in pregnancy in Kenya: design, methods, and baseline results of a cluster-randomized controlled trial. PLoS One. 2012;7(9):e44181. doi: 10.1371/journal.pone.0044181. Epub 2012 Sep 6. PMID 22970177